CLINICAL TRIAL: NCT00695045
Title: Determination of the Efficacy and Side-Effect Profile of Lower Doses of Intrathecal Morphine in Patients Undergoing Total Knee Arthroplasty
Brief Title: Intrathecal Morphine in Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Hospital Galway (Other)
Responsible Party: Dr Patrick Hassett, Department of Anaesthesia , University College Hospital Galway
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2008-06-11 (Estimated); Status verified 2008-06

CONDITIONS: Pain, Postoperative; Arthroplasty, Replacement, Knee
Keywords: Pain, Postoperative; Arthroplasty, Replacement, Knee; Morphine; Injections, Intrathecal
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): patients in this group got 100mcg of intrathecal morphine.
  Interventions: Drug: intra thecal morphine
- 2 (Experimental): patients in this group got 200 mcg intrathecal morphine
  Interventions: Drug: intra thecal morphine
- 3 (Experimental): patients in this group given 300 mcg intrathecal morphine.
  Interventions: Drug: intra thecal morphine

INTERVENTIONS:
Drug: intra thecal morphine — 100 mcg intrathecal morphine given once .
  Other Names: intraspinal morphine
  Arms: 1
Drug: intra thecal morphine — 200 mcg intrathecal morphine given once
  Other Names: intra spinal morphine
  Arms: 2
Drug: intra thecal morphine — 300 mcg intrathecal morphine given once
  Other Names: intra spinal morphine
  Arms: 3

SUMMARY:
This study is designed to explore the efficacy lower doses of intra-spinal morphine for pain relief and side effect profiles of same in the setting of Total Knee Replacement.We hypothesized that a dose greater than that used in Total Hip Replacement was needed and wished to find a dose which was effective but had a low side effect profile.

ELIGIBILITY:
Inclusion Criteria:

* Patients for elective total knee arthroplasty

Exclusion Criteria:

* No contraindication to spinal
* No allergy to morphine, rescue analgesia or anti-emesis treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-07; Primary Completion 2007-01 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
pain | 24 hours

SECONDARY OUTCOMES:
nausea and vomiting | 24 hours
pruritus | 24 hours
sedation | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Patrick D Hassett, MD, Principal Investigator — Department of Anaesthesia, UCHG; John Laffey, MD, Study Chair — Department of Anaesthesia,UCHG; Brian Kinirons, MD, Study Director — Dept of Anaesthesia , UCHG

REFERENCES:
- [Derived] Hassett P, Ansari B, Gnanamoorthy P, Kinirons B, Laffey JG. Determination Of The Efficacy And Side-effect Profile Of Lower Doses Of Intrathecal Morphine In Patients Undergoing Total Knee Arthroplasty. BMC Anesthesiol. 2008 Sep 24;8:5. doi: 10.1186/1471-2253-8-5. PMID 18816386